CLINICAL TRIAL: NCT05394103
Title: A Phase 1/2 Multicenter, Open-label, Dose-escalation, Safety, Pharmacodynamic, and Pharmacokinetic Study of Q901Administered Via Intravenous Infusion as Monotherapy and in Combination With Pembrolizumab in Adult Patients With Selected Advanced Solid Tumors With Cohort Expansions at the Recommended Phase 2 Dose
Brief Title: Highly Selective CDK7 Inhibitor Q901 in Selected Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qurient Co., Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QRNT-009; MK-3475-E45 (KEYNOTE-E45) (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation (Q901) (Experimental)
  Interventions: Drug: Q901
- Q901 Single-Agent Expansion Cohorts (Experimental)
  Interventions: Drug: Q901
- Q901 + KEYTRUDA® (pembrolizumab) Cohorts (Experimental)
  Interventions: Drug: Q901; Drug: KEYTRUDA® (pembrolizumab)

INTERVENTIONS:
Drug: Q901 — The study drug Q901 will be administered by IV infusion over a 30-minute period using a QW dosing schedule for 4 weeks, followed by a Q2W interval dosing schedule thereafter
Drug: KEYTRUDA® (pembrolizumab) — KEYTRUDA® (pembrolizumab) will be administered Q6W
  Arms: Q901 + KEYTRUDA® (pembrolizumab) Cohorts

SUMMARY:
Multicenter, open-label, dose-escalation, safety, tolerability, PK and pharmacodynamic study with a dose expansion at the RP2D to evaluate safety and potential antitumor activity of Q901 as a monotherapy and in combination with pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed advanced or metastatic ovarian, CRPC, HR+ HER2- breast, endometrial, colorectal, small-cell lung, or pancreatic cancer, who have progressed following standard-of-care therapy or for whom there is no standard therapy that confers clinical benefit
* Measurable disease per RECIST v 1.1
* ECOG performance status 0,1 or 2
* Life expectancy of at least 3 months
* Age ≥ 18 years
* Signed, written IRB-approved informed consent form

Exclusion Criteria:

* New York Heart Association Class III or IV cardiac disease, or myocardial infarction, severe unstable angina, coronary/peripheral artery bypass graft, congestive heart failure within the past 6 months
* Have a corrected QT interval (using Fridericia's correction formula) (QTcF) of >470 msec (females) and >450 msec (males)
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Active, poorly controlled autoimmune or inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 28 days of cycle 1 (each cycle is 28 days)

SECONDARY OUTCOMES:
Change in the area under curve (AUC) of Q901 | Cycle 1 Day 1 and Day 22, Cycle 2 Day 8 and Day 22 (each cycle is 28 days)
Change in the maximum plasma concentration (Cmax) of Q901 | Cycle 1 Day 1 and Day 22, Cycle 2 Day 8 and Day 22 (each cycle is 28 days)
Change in the time of maximum plasma concentration (Tmax) of Q901 | Cycle 1 Day 1 and Day 22, Cycle 2 Day 8 and Day 22 (each cycle is 28 days)
Tumor response using RECIST version 1.1 throughout study | Baseline and at the end of every even cycle up to approximately 2 years (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - Mayo Clinic, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Atlantic Health System Hospital, Morristown, New Jersey
  - Mary Crowley Cancer Research, Dallas, Texas
- South Korea (4):
  - National Cancer Center, Goyang-si
  - CHA University Bundang Medical Center, Seongnam-si
  - Asan Medical Center, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided